CLINICAL TRIAL: NCT03529188
Title: Validation of the French Version of the Three Scales for Assessing the Fear of Type 1 Hypoglycemia (HFS-C, HFS-PYC and HFS-P) in Children, Adolescents and Their Parents by a Monocentric Transverse Psychometric Study
Brief Title: French Version of the Scales of Fear of Hypoglycaemia in Children With Type 1 Diabetes and Their Parents
Acronym: FHS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: FOH (29BRC17.0161)
Record Dates: First submitted 2018-03-13; First posted 2018-05-18 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Type 1
Keywords: Diabetes type 1; Child ans teenager; Fear of Hypoglycaemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Type 1 diabetes usually appears brutally in children or young adults. While many factors of poor glycemic balance have been identified in the literature (age, socio-cultural and socio-economic level, family structure, adherence etc.), it turns out that hypoglycemia is the most common acute complications. It would be an important physiological and psychological barrier for the patient and his parents to manage this diabetes, the latter seeking to keep the blood glucose levels above the objectives in order to avoid the occurrence of a hypoglycemia, especially nocturnal.

If there is a questionnaire currently validated as a tool to measure the fear of hypoglycemia (HFS, Hypoglycemia Fear Survey is available in three versions: L'HFS-Child (HFS-C) for children over 6 years old, HFS-Parents of Young children ( HFS-PYC) for parents of young children (under 8 years of age) and HFS-Parents (HFS-P)) for parents of children over 8 years of age, on the other hand, there are no French and no French studies have evaluated the prevalence and impact of the fear of hypoglycemia in French patients with type 1 diabetes.

It is therefore essential to use a reliable and valid tool to identify patients affected by the fear of hypoglycemia, which can be an obstacle to improve glycemic control and to an optimum quality of life. Having a tool in French and validated on the scientific level would allow to propose adapted therapeutic treatments (psychological follow-up, individual or collective sessions of therapeutic education, material assistance (sensor of blood glucose, pump with insulin stop...) In order to both improve metabolic balance while increasing the quality of life of patients by lowering secondary anxiety to hypoglycemia

ELIGIBILITY:
Inclusion Criteria:

* Age between 2 and 18 years
* Type 1 diabetes defined by an hyperglycemia higher than 2g/l, polyuria, polydipsia and positive antibody
* insulin-treated type 2 diabetes by daily injections or insulin pump

Exclusion Criteria:

* Trouble to read
* Trouble to understand
* Trouble to answer to the questionnaire
* Opposition.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — male or female
Study Population: Child and teenager with Type 1 diabetes defined by an hyperglycemia higher than 2g/l, polyuria, polydipsia and positive antibody.
Sampling Method: Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2018-08-03 (Actual); Primary Completion 2020-12-03 (Estimated); Study Completion 2020-12-03 (Estimated)

PRIMARY OUTCOMES:
HFS-Child score, | Month 0
  Change of Behaviour adopted by the patient in order to avoid the occurrence of hypoglycemia and worry about low blood sugar
HFS-PYC score | Month 0, Month 3 (+/- 30 days)
  Change in Anxiety related to the phenomenon of hypoglycemia
HFS-Parent score | Month 0, Month 3 (+/- 30 days)
  Change of Behaviour adopted by the parent in order to avoid the occurrence of hypoglycemia

SECONDARY OUTCOMES:
Questionnaire Survey "children " | Month 0, Month 3 (+/- 30 days)
  Diabetes impact on relationships, activity, alimentation ... " children"
Questionnaire Survey "parents " | Month 0, Month 3 (+/- 30 days)
  Diabetes impact on relationships, activity, alimentation ... " parents"
HbA1C | Month 0, Month 3 (+/- 30 days)
  percentage value

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHRU de Brest, Brest
  - Centre Hospitalier de Bretagne Sud, Lorient
  - Hôpital Universitaire Robert-Debré, Paris

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending three years maximum following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. requestors will be required to sign and complete a data access agreement